CLINICAL TRIAL: NCT05676970
Title: Using a Telehealth and Shared Decision-Making Model to Address Preventative Medicine Strategies Among Communities in Louisiana
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xavier University of Louisiana. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB938-24
Record Dates: First submitted 2022-12-19; First posted 2023-01-09 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Preventative Medicine
Keywords: Diabetes; Hypertension; Hyperlipidemia; Medication Compliance; Nutrition; Exercise
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias; Medication Adherence; Motor Activity

STUDY DESIGN:
Intervention Model Description: We propose to use a individually randomized group treatment trial design with a baseline survey to assess social determinants of health, baseline demographic information and preventive medicine strategies. We will then randomize participants in a 1:1 fashion to a personalized preventative medicine intervention arm and a control arm. Given this is an IRGT (Individualized Randomized Group Treatment) trial design, a priori matching should assist in preventing a Type I error. Individuals will then complete 5 individual or group based behavioral health interventions via a Telehealth model conducted by a Clinical Pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telehealth Arm: Personalized Preventative Medicine Strategies (Experimental): Individuals in this arm will complete a personalized telehealth interventions that focus on nutrition, work-life balance, medication compliance, herbals, exercise targets hyperlipidemia, diabetes and hypertension around individual risks for development of the disease state. All educations will be completed one-on-one as well as small group.
  Interventions: Behavioral: Telehealth: Personalized Preventative Medicine Strategies
- Telehealth Arm: Preventative Medicine Education (Active Comparator): Individuals in this arm will complete standardized telehealth interventions that focus on nutrition, work-life balance, mental health, diabetes and hypertension general education. All educations will be completed one-on-one as well as small group.
  Interventions: Behavioral: TeleHealth: Preventative Medicine Education

INTERVENTIONS:
Behavioral: Telehealth: Personalized Preventative Medicine Strategies — Individuals in this arm will complete a personalized telehealth interventions that focus on nutrition, work-life balance, medication compliance, herbals, exercise targets hyperlipidemia, diabetes and hypertension around individual risks for development of the disease state. All educations will be completed one-on-one as well as small group.
  Arms: Telehealth Arm: Personalized Preventative Medicine Strategies
Behavioral: TeleHealth: Preventative Medicine Education — Individuals in this arm will complete standardized telehealth interventions that focus on nutrition, work-life balance, mental health, diabetes and hypertension general education. All educations will be completed one-on-one as well as small group.
  Arms: Telehealth Arm: Preventative Medicine Education

SUMMARY:
This study is a 12-18 month behavioral intervention study to assess the impact of enrolling individuals a clinical pharmacist run Telehealth education focused on wellness and preventive health strategies. Individuals will be randomized to either a wellness education only model focusing on nutrition, diabetes, hyperlipidemia and hypertension or a wellness education model with personalized preventative medicine strategies for the patient. All participants will complete individual and group based interventions. Individuals will be recruited from target work industries such as health workers, teachers aides and the food industry. We are recruiting individuals who come from urban, semi-rural or rural communities or have additional social determinants of health that indicate social vulnerability. The primary outcome is willingness to participate in preventative medicine strategies to prevent development of chronic medical conditions. The secondary outcome is barriers to preventive medicine strategies including for chronic preventable disease such as nutrition, hypertension, hyperlipidemia, diabetes and medication compliance.

DETAILED DESCRIPTION:
Individuals will be recruited using a community-based participatory research model to identify 360 patients to enter into an 12-18 month clinical pharmacist run, preventative medicine strategies including; health and wellness program delivered via Xavier's clinical pharmacy faculty trained in telehealth medicine using an individually randomized group treatment trial approach based upon industry of recruitment. Participants will be recruited from target high risk industries for respiratory infection: hospitality and food industry, plant workers, nurse's aides, teacher's aides and the beauty industries. Participants will complete a minimum of three individual visits and group informational visits with a target of five sessions total. Both arms of the study will receive health and wellness education around target topics of diabetes, hypertension, hyperlipidemia, nutrition, exercise, herbals and medication compliance. Only the preventative medicine education intervention arm will receive the preventative medicine education including personalized counseling around the target disease states, medication reviews, medication-nutrition reviews and development of a personalized plan. Measures in changes in preventative health behaviors will occur by the clinical pharmacist via patient interviews. The primary outcome will be preventative medicine strategies knowledge preventable chronic diseases such as diabetes, hypertension and hyperlipidemia. The secondary outcome will be assessing barriers for preventive health behaviors.

Impact: The implications of this proposed project are to understand health related beliefs and behaviors related to preventative medicine strategies in the context of a general health and wellness model.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years to 55 years of age
2. Able to speak English
3. Currently employed or seeking training in target industries such as: healthcare, education, beauty, hospitality, food (culinary) and industrial plant workers.
4. Able to use Telehealth technology via tablet, cell phone, or computer

Exclusion Criteria:

1. Individuals who are unable to give informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Willingness to participate in preventative medicine screening for Diabetes, Hypertension and Hyperlipidemia | 12 months, completed year 1 of the study.
  Questionnaire derived from Documented preventative medicine strategies; Ordinal Variable: Scale of 1 to 5 (Least Likely to Most Likely)
Participating in Screening for DM, hypertension, hyperlipidemia | Through study completion, on average, 12-18 months
  Participated in preventative medicine screening activity such as fasting blood glucose, blood pressure check and lipid panels. Binary Variable: Yes or No
Willingness to participate in personalized exercise and nutrition goals to prevent chronic disease | Through study completion, on average, 12-18 months
  Questionnaire derived from Documented preventative medicine strategies; Ordinal Variable: Scale of 1 to 5 (Least Likely to Most Likely)
Participating in personalized exercise and nutrition goals | Monthly through study completion, on average, 12-18 months
  After development of personalized exercise and nutrition goals with Telehealth pharmacist, documented participation in activities at least once per week. Data will be recorded monthly as a Binary Variable: Yes or No
Participating in personalized medication compliance for prescription, over the counter, herbals and nutraceuticals related to health promotion | Monthly through study completion, on average, 12-18 months
  After development of personalized exercise and nutrition goals with Telehealth pharmacist, documented participation in activities at least once per week. Data will be recorded monthly as a Binary Variable: Yes or No

SECONDARY OUTCOMES:
Barriers to preventative medicine strategies | Through study completion, on average, 12-18 months
  Work place barriers will be assessed as dichotomized variables such as: insurance access, paid time off for illness, work schedules consistent permitting medical appointments, and medication compliance.
Knowledge of personal disease risk (diabetes, hypertension, hyperlipidemia) using standardized education tools | Baseline, after corresponding session, end of program: Through study completion, on average, 12-18 months
  10 question knowledge test, Scored as minimally competent at 70% correct, scored as binary
Knowledge of risk factors and personal risk for diabetes, hypertension and hyperlipidemia | Baseline, after corresponding session, end of program: Through study completion, on average, 12-18 months
  10 question knowledge test, Scored as minimally competent at 70% correct, scored as binary
Knowledge of personalized medication compliance for prescription, over the counter, herbals and nutraceuticals related to health promotion | Baseline, after corresponding session, end of program: Through study completion, on average, 12-18 months
  10 question knowledge test, Scored as minimally competent at 70% correct, scored as binary

CONTACTS AND LOCATIONS:
Overall Officials: Sara Al-Dahir, PhD, Principal Investigator — Xavier University of Louisiana.; Klaus Heyer, PhD, Principal Investigator — Nunez Community College
Locations (1):
- Xavier University of Louisiana, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request, we will share our intervention and information below.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of study.
Access Criteria: Approval by Principal Investigator.
URL: http://www.xulavoice.com/telehealth